CLINICAL TRIAL: NCT00447668
Title: Effect of Yoga Vs. Stretching on Chronic Back Pain
Acronym: YES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01AT003208 (NIH); U01AT003208 (NIH)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Chronic Low Back Pain; Yoga
MeSH Terms: interventions — Yoga; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Yoga
- 2 (Active Comparator): Exercise
  Interventions: Behavioral: Exercise
- 3 (Active Comparator): Self-care book recommendations
  Interventions: Behavioral: Self-care book recommendations

INTERVENTIONS:
Behavioral: Yoga — Yoga for back pain
  Arms: 1
Behavioral: Exercise — exercises for back pain
  Arms: 2
Behavioral: Self-care book recommendations — Self-care book for back pain
  Arms: 3

SUMMARY:
This study will compare the effectiveness of yoga classes, exercise classes, and a self-care book in the management of pain and function for people with low back pain.It will also for physical, psychological and physiological factors associated with improvement in back pain.

ELIGIBILITY:
Inclusion Criteria:

* Group Health Cooperative enrollee
* Uncomplicated low back pain
* At least moderate pain levels

Exclusion Criteria:

* Sciatica persisting 3 or more months after physician visit
* History of cancer (other than nonmelanoma skin cancer)
* Severe disk problems
* Unstable medical conditions
* Back surgery within past 3 years
* Physically unable to do the yoga or exercise classes and homework
* Unable to attend classes
* Currently doing yoga
* Taken yoga or exercise class for back pain within past year
* Currently in litigation for back pain
* Seeking other treatment for back pain

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Back-related function | 6 months
Pain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Sherman, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Sherman KJ, Cherkin DC, Wellman RD, Cook AJ, Hawkes RJ, Delaney K, Deyo RA. A randomized trial comparing yoga, stretching, and a self-care book for chronic low back pain. Arch Intern Med. 2011 Dec 12;171(22):2019-26. doi: 10.1001/archinternmed.2011.524. Epub 2011 Oct 24. PMID 22025101
- [Derived] Sherman KJ, Cherkin DC, Cook AJ, Hawkes RJ, Deyo RA, Wellman R, Khalsa PS. Comparison of yoga versus stretching for chronic low back pain: protocol for the Yoga Exercise Self-care (YES) trial. Trials. 2010 Mar 31;11:36. doi: 10.1186/1745-6215-11-36. PMID 20356395